CLINICAL TRIAL: NCT00394823
Title: A Randomized, Open-label, Multicentric Parallel Group Study to Assess the Impact of Supportive Measures on the Drug Adherence of Patients With Essential Hypertension Treated With Valsartan or Valsartan Plus HCTZ for 34 Weeks With or Without Respective Measures
Brief Title: VALIDATE Valsartan and Supportive Measures - Impact on Drug Adherence of Treated Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CVAL489ADE24
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
Keywords: Hypertension, valsartan, compliance
MeSH Terms: conditions — Hypertension; Patient Compliance

INTERVENTIONS:
Behavioral: Set of supportive tools/measures vs. standard care

SUMMARY:
The purpose of this study is to assess the impact of supportive measures on the drug adherence of patients with essential hypertension

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients >= 18 years
* Females must be either post-menopausal for one year, surgically sterile or using effective contraceptive methods (e.g. barrier method with spermicide, intra-uterine device, hormonal contraceptives).
* Patients with mild essential hypertension: Systolic blood pressure ≥ 140 mmHg and < 170 and/or diastolic blood pressure ≥ 90 mmHg and < 105 mmHg"

Exclusion Criteria:

* Moderate and severe hypertension
* Pregnant or nursing women
* A history of cardiovascular disease, including angina pectoris, myocardial infarction, coronary artery bypass graft, percutaneous transluminal coronary angioplasty, transient ischemic attack, stroke, and heart failure NYHA II - IV

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2005-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Drug adherence in patients (daily proportion of patients taking one tablet of the prescribed hypertensive therapy as prescribed)

SECONDARY OUTCOMES:
Compliance and persistence between randomized groups over time.
To assess discrepancies between pill counts, Morisky questionnaire and electronic monitoring to estimate patient adherence to prescribed therapy
To assess the relation between drug exposure and BP reduction.
To assess the relation between drug exposure and the likelihood to switch to valsartan 160 mg plus HCTZ 12.5 mg
To assess the safety and tolerability of valsartan 160 mg and valsartan 160 mg plus
HCTZ 12.5 mg.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Basel, Study Chair — +41 61 324 1111
Locations (2):
- Investigative Centers, Germany
- Novartis, Basel, Switzerland

REFERENCES:
- [Derived] Dusing R, Handrock R, Klebs S, Tousset E, Vrijens B. Impact of supportive measures on drug adherence in patients with essential hypertension treated with valsartan: the randomized, open-label, parallel group study VALIDATE. J Hypertens. 2009 Apr;27(4):894-901. doi: 10.1097/HJH.0b013e328323f9be. PMID 19300114